CLINICAL TRIAL: NCT06550258
Title: Effects of Hippotherapy on Upper Extremity Functionality and Trunk Control in Children With Cerebral Palsy
Brief Title: Effects of Hippotherapy on Functionality in Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, tuba kolaylı, Lecturer, Uskudar University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 61351342/2019-399
Record Dates: First submitted 2024-08-05; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Palsy
Keywords: hippotherapy; physiotherapy; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Before - after trial
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hippotherapy group (Experimental): Hippotherapy was applied with a physiotherapist for 2 months.
  Interventions: Other: Equine-assisted therapy
- Control group (Active Comparator): Classical physiotherapy was applied with the help of a physiotherapist for 2 months.
  Interventions: Other: Traditional Pediatric Physiotherapy

INTERVENTIONS:
Other: Equine-assisted therapy — Hippotherapy is a therapeutic intervention applied by physiotherapists that aims to improve impaired body functions. Hippotherapy is a therapy in which the rider receives stimuli from the horse that stimulate the sensory, neuromotor and cognitive systems during riding and exercise on the back of a horse. Hippotherapy is effective on posture control, balance, gross motor functions and functional performance in children with cerebral palsy.
  Arms: Hippotherapy group
Other: Traditional Pediatric Physiotherapy — In traditional pediatric physiotherapy, cushions of appropriate hardness were used for proprioceptive input. Stools of different heights were used for sitting, squatting, standing up by holding on and standing, Bobath balls and balance boards were used for balance reactions. Triangular and roll cushions of different hardness were used for weight transfer. Surfaces with different patterns were used for sensory input. The child's wishes and interests were taken into consideration in the selection of materials. The treatment was planned according to the activities that were difficult in daily life and the aim was to transfer the knowledge learned to daily life.
  Arms: Control group

SUMMARY:
The purpose of this clinical review is to investigate the effect of hippotherapy in improving upper limb functionality in children with cerebral palsy. The main question it aims to answer is The questions are as follows:

1. Does hippotherapy improve gross motor function of the upper extremity in children with cerebral palsy?
2. Is the development of trunk control in children with cerebral palsy who receive hippotherapy different from the development of trunk control in children who receive conventional physiotherapy?

Participants will:

Hippotherapy and routine physiotherapy in 2 different groups for 2 They will carry out the necessary evaluations before the implementation and at the end of 2 months.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a permanent developmental disorder that occurs as a result of a lesion in the developing baby's brain. Due to the symptoms seen in CP, the individual's participation in daily living activities (ADL) is restricted and functional mobility is affected. Hippotherapy is preferred in children with CP because it includes fun activities and is effective in terms of the child's participation and motivation. The aim of this study is to examine the effect of hippotherapy on upper extremity function. In this study planned as a multicenter study, children with CP are divided into 2 groups as the study and control groups. After a 2-month application, children with CP will be evaluated in terms of upper extremity functionality and postural control. The "Statistical Package for Social Sciences (SPSS) Statistics 23.0 (SPSS Inc, Chicago, USA) program will be used in the analysis of the study data. The change in numerical variables over time in the treatment and control groups and the group-time interaction will be examined with "two-way repeated measures variance analysis". The "Chi-Square Test" will be used to examine the relationship between categorical variables. The relationship between numerical variables will be examined with the "Spearman rho correlation coefficient". The probability of error will be accepted as (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with SP
* Being between the ages of 4-16
* Being at GMFCS (Gross Motor Function Classification System) level 1,2 or 3
* Being at MACS (The Manual Ability Classification System) level 1,2,3 or 4
* Having a stable clinical condition
* Having the cognitive level to follow the instructions in the test and treatment protocol

Exclusion Criteria:

* Families who do not sign the consent form
* Presence of active seizures
* Presence of developmental hip dysplasia
* Presence of allergy to horses
* Having undergone surgical intervention or Botulinum Toxin A (BTX-A) application in the last 6 months

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Box and block test | 8 weeks
  This test evaluates manual dexterity. The person being tested is asked to move blocks from one compartment to the other compartment as fast as they can within 60 seconds. The test is started with the dominant hand and the test is repeated with both hands. In addition, a 15-second trial period is given for both hands. The blocks are held in the compartment on the side of the hand to be tested, and the test is started by positioning the box in the midline of the person being tested. When the time is up, the blocks carried are counted and the result is recorded.
Trunk Control Measurement Scale | 8 weeks
  The Trunk Control Measurement Scale includes 15 items that measure the two main components of trunk control, static and dynamic sitting balance. The Static Sitting Balance Scale (items 1-5) evaluates the ability to maintain stable trunk posture during movements of the upper and lower extremities. The Dynamic Sitting Balance Scale (items 6-15) is divided into two subscales: the selective movement control scale and the dynamic reach scale. The total score ranges from 0-58. A high score indicates good performance.

SECONDARY OUTCOMES:
ABILHAND-Kids | 8 weeks
  It is used to measure hand functions in children with CP. It aims to measure the use of the upper extremity in children's daily activities in 21 items (It is examined in 3 columns as cannot be done, difficult, easy. It mostly evaluates the function of both hands together. The scale is generally applied by asking the families, if the child is older, he/she can be included in the application. There should be no assistive device or human support while evaluating the functional ability.
Moberg pickup test | 8 weeks
  In a performance-based (timed) manual dexterity test, the patient is asked to fill certain items into a box. The test is started with the dominant hand, then with the non-dominant hand and with eyes closed. The test is repeated 3 times and the best time on the stopwatch is noted.
Gross Motor Function Measure | 8 weeks
  GMFM-88 is a scale developed for children with CP to show changes in gross motor functions. It is divided into 5 main sections as lying-rolling, sitting, crawling-kneeling, standing, walking-running-jumping. The values are divided into 4 categories as -Cannot initiate the activity ''0'', -Initiates independently ''1'', -Partially completes ''2'', -Completes independently ''3''. The total score is calculated as a percentage, as the percentage values increase, motor functions increase.

CONTACTS AND LOCATIONS:
Locations (1):
- Uskudar University, Istanbul, Ümraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Champagne D, Corriveau H, Dugas C. Effect of Hippotherapy on Motor Proficiency and Function in Children with Cerebral Palsy Who Walk. Phys Occup Ther Pediatr. 2017 Feb;37(1):51-63. doi: 10.3109/01942638.2015.1129386. Epub 2016 Mar 1. PMID 26930110
- [Background] Park ES, Rha DW, Shin JS, Kim S, Jung S. Effects of hippotherapy on gross motor function and functional performance of children with cerebral palsy. Yonsei Med J. 2014 Nov;55(6):1736-42. doi: 10.3349/ymj.2014.55.6.1736. PMID 25323914
- [Background] Kwon JY, Chang HJ, Yi SH, Lee JY, Shin HY, Kim YH. Effect of hippotherapy on gross motor function in children with cerebral palsy: a randomized controlled trial. J Altern Complement Med. 2015 Jan;21(1):15-21. doi: 10.1089/acm.2014.0021. Epub 2014 Dec 31. PMID 25551626